CLINICAL TRIAL: NCT05411029
Title: Disrupted Sleep in Somali Americans - Implications for Hypertension Risk
Brief Title: Study of Disrupted Sleep in Somali Americans
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Virend Somers, MD, PhD, Principal Investigator, Mayo Clinic
Other Study IDs: 22-004192
Record Dates: First submitted 2022-06-06; First posted 2022-06-08 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Hypertension; Sleep Disorder; Healthy
MeSH Terms: conditions — Hypertension; Sleep Wake Disorders | interventions — Blood Pressure; Polysomnography

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Somali Americans: Somali Americans with no known history of hypertension, diabetes, or sleep disorders will have a 24 hour blood pressure monitoring and polysomnography.
  Interventions: Diagnostic Test: 24 hour blood pressure (BP) monitoring; Diagnostic Test: Polysomnography

INTERVENTIONS:
Diagnostic Test: 24 hour blood pressure (BP) monitoring — 24-hour ambulatory BP measuring device and blood pressures will be measured every 20 minutes to half hour
Diagnostic Test: Polysomnography — Measurements will include electroencephalogram, electromyogram, electrooculogram, electrocardiogram, breathing patterns of chest and abdomen, nasal and oral airflow and oxygen saturation. Sleep stages and apneas will be scored in accordance with validated American Academy of Sleep Medicine standards.
  Other Names: Sleep Study

SUMMARY:
The aims of this study are to determine the types and severity of previously undiagnosed sleep deficiencies in otherwise healthy Somali Americans, apply a research framework to define psychosocial, behavioral, environmental, and biological mechanisms mediating sleep deficiencies in Somali Americans, and examine the relationship between sleep deficiencies and increased blood pressure in Somali Americans.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with no known history of hypertension, diabetes, or sleep disorders.
* Self-identify as Somali.
* Adult males and females who are older than 18 years of age.

Exclusion Criteria:

* Anyone under 18 years or over 70 years.
* Positive pregnancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The research team will partner with Somali operated community-based health clinics, faith-based establishments, community organizations, charter schools and other educational/community centers. In addition, the research team will partner with the Somali Health Advisory Committee (SHAC), a community advisory board based in Rochester and Minneapolis/St. Paul and the Somali Community Resettlement Agency (SCRS) and Somali American Social Services Association (SASSA), two community organizations aimed at integrating Somali immigrants to the United States.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Undiagnosed sleep deficiency-short sleep | 1 night sleep study, approximately 8-9 hours
  Number of subjects to have short sleep (<6 hours) as measured by the sleep study
Undiagnosed sleep deficiency-insomnia | 1 night sleep study, approximately 8-9 hours
  Number of subjects to have insomnia as measured by the sleep study
Undiagnosed sleep deficiency-obstructive sleep apnea (OSA) | 1 night sleep study, approximately 8-9 hours
  Number of subjects to have OSA as measured by the sleep study
Disrupted sleep | 1 night sleep study, approximately 8-9 hours
  Number of subjects to have disrupted sleep as measured by the sleep study
Blood pressure (BP) during wakefulness | Day 2
  Average BP as measured by 24 hour BP monitoring, reported in mmHg
Blood pressure (BP) during sleep | Day 2
  Average BP as measured by 24 hour BP monitoring, reported in mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Virend Somers, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Greenlund IM, Bock JM, Govindan N, Kantas D, Singh P, Covassin N, Somers VK. Blood Pressure and Heart Rate Response to Orthostasis in Somali Americans. J Racial Ethn Health Disparities. 2025 Mar 15:10.1007/s40615-025-02389-7. doi: 10.1007/s40615-025-02389-7. Online ahead of print. PMID 40088388
- [Derived] Greenlund I, Bock J, Govindan N, Kantas D, Singh P, Covassin N, Somers V. Blood Pressure and Heart Rate Response to Orthostasis in Somali Americans. Res Sq [Preprint]. 2024 Oct 21:rs.3.rs-4925722. doi: 10.21203/rs.3.rs-4925722/v1. PMID 39502777